CLINICAL TRIAL: NCT00335036
Title: Pediatric Lead Extractability and Survival Evaluation (PLEASE)Study: A Prospective Assessment of Implantable Cardioverter Defibrillator (ICD) Lead Extractability and Survival in Children and Congenital Heart Disease Patients
Brief Title: Pediatric Lead Extractability and Survival Evaluation (PLEASE)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lead was recalled and manufacturing halted
Sponsor: Elena Gibson (Other)
Collaborators: Medtronic (Industry); Guidant Corporation (Industry)
Responsible Party: Sponsor-Investigator, Elena Gibson, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHB-05-11-147
Record Dates: First submitted 2006-06-06; First posted 2006-06-08 (Estimated); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation; Cardiomyopathy; Long QT Syndrome; Congenital Heart Disease
Keywords: Implantable Cardioverter Defibrillator; Ventricular Arrhythmia; Sudden Cardiac Death; Congenital Heart Disease; Pediatric Electrophysiology
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Cardiomyopathies; Long QT Syndrome; Heart Defects, Congenital; Death, Sudden, Cardiac

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thin leads (Active Comparator): Thin (less than or equal to 7 French introducer) isodiametric ICD leads
  Interventions: Device: Thin leads
- Gore PTFE-coated (Active Comparator): ICD lead with PTFE-coated coils
  Interventions: Device: ICD lead implant

INTERVENTIONS:
Device: ICD lead implant — Randomization of ICD lead type at implant
  Arms: Gore PTFE-coated
Device: Thin leads — Thin (less than or equal to 7 French introducer) isodiametric ICD leads
  Arms: Thin leads

SUMMARY:
This is a randomized, prospective clinical trial comparing 2 different types of implantable cardioverter defibrillator (ICD) leads in children and patients with congenital heart disease. ICD lead survival in this patient group is particularly suboptimal, and lead extraction is technically difficult and carries a substantial morbidity risk. Recently, improved ICD lead designs have been released and are currently being utilized in patients. The main aim of the study is to determine if either type of lead performs better in terms of implantation electrical characteristics, long-term survival without breaking, and ease of extractability.

DETAILED DESCRIPTION:
The recognition that ICD therapy in children can be life-saving, as well as the development of smaller devices and leads, are resulting in increased ICD implantation in the pediatric and young adult populations. However, ICD lead survival in this patient group is suboptimal. Lead extraction is technically difficult and has substantial morbidity. Recently, improved ICD lead designs have been released and are currently being utilized. While the development of transvenous ICD leads has allowed for less invasive implantation, the long-term presence of these leads carries some risks. When a lead becomes infected or causes patient morbidity, it must be removed. Because of the larger caliber of ICD leads and the presence of uninsulated shocking coils, non-functional ICD leads usually warrant removal to avoid future mechanical or electrical lead interactions. The larger size of ICD leads is of concern in this younger population, particularly with regard to avoiding the accumulation of implanted hardware. The principal indication for lead revision in children and young adults is lead malfunction, commonly related to patient growth and increased physical activity in this younger population. The removal of chronic indwelling pacer or ICD leads is not trivial. Scar tissue begins to bind transvenous leads to the endothelial surface several weeks after implantation, and this fibrous adherence progresses over time, exacerbated by high-energy shock delivery. In children and younger adult ICD recipients, exuberant lead scarring is prevalent, particularly in the regions of venous entry, high voltage shocking coils, and the lead tip. Transvenous lead extraction has been facilitated by the use of telescoping sheaths and powered sheaths that can be advanced over the lead to disrupt scar tissue and free the lead from the endothelium.

The 2 ICD lead types to be compared (thin ICD leads versus ePTFE-coated leads) in the proposed study are at clinical equipoise. Both types are believed to be improved over prior generation ICD leads. However, a direct comparison has not been performed. As the pediatric and congenital heart disease patient subgroup is younger than the average ICD patient population, they will have greater likelihood of long-term survival, and therefore, the issues of lead survival, durability, and extractability are critically important. While these themes are important for all ICD patients, they are particularly germane for younger patients who have more active lifestyles and are, in general, expected to outlive their ICD leads.

This study will prospectively assess the improvements in ICD lead design, specifically comparing a Gore ePTFE coating and thinner caliber ICD leads in pediatric and congenital heart disease population.

Specific Aim #1: To prospectively evaluate the long-term performance of modern-generation ICD leads in pediatric and congenital heart disease patients.

Specific Aim #2: To determine the potential beneficial effects of two improvements in ICD lead design - Gore ePTFE coil coating and thinner lead diameter in pediatric and congenital heart disease patients.

Specific Aim #3: To directly compare the safety and efficacy of these new ICD lead technologies in terms of extractability in pediatric and congenital heart disease patients.

The primary hypothesis is that improved lead designs and smaller diameter leads will demonstrate benefit in survival and extractability. The primary outcome variables will include: a) ICD lead functionality and performance by subtype, b) inappropriate shocks due to lead issues, c) lead extractability by subtype (Gore-coated versus thin leads).

Secondary outcomes include comparison of implant electrical parameters, patient morbidity and mortality, comparing each new lead type with each other and against historical pediatric controls with standard transvenous ICD leads.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for study enrollment at the time of implantation of a new ICD and transvenous ICD lead.
* All patients under the age of 21 years at the time of initial ICD implantation, or those patients with congenital heart disease and an indication for ICD implantation are eligible for participation.

Exclusion Criteria:

* Patients who have existing ICD leads in place.
* Patients with expected survival less than 1 year.
* Patients who cannot be expected to participate in follow-up visits.
* Patients receiving an epicardial or subcutaneous ICD (without transvenous ICD lead).

Ages: 1 Year to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 748 (Actual)
Dates: Start 2006-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles I Berul, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Alexander ME, Cecchin F, Walsh EP, Triedman JK, Bevilacqua LM, Berul CI. Implications of implantable cardioverter defibrillator therapy in congenital heart disease and pediatrics. J Cardiovasc Electrophysiol. 2004 Jan;15(1):72-6. doi: 10.1046/j.1540-8167.2004.03388.x. PMID 15028076
- [Background] Stephenson EA, Batra AS, Knilans TK, Gow RM, Gradaus R, Balaji S, Dubin AM, Rhee EK, Ro PS, Thogersen AM, Cecchin F, Triedman JK, Walsh EP, Berul CI. A multicenter experience with novel implantable cardioverter defibrillator configurations in the pediatric and congenital heart disease population. J Cardiovasc Electrophysiol. 2006 Jan;17(1):41-6. doi: 10.1111/j.1540-8167.2005.00271.x. PMID 16426398
- [Background] Cooper JM, Stephenson EA, Berul CI, Walsh EP, Epstein LM. Implantable cardioverter defibrillator lead complications and laser extraction in children and young adults with congenital heart disease: implications for implantation and management. J Cardiovasc Electrophysiol. 2003 Apr;14(4):344-9. doi: 10.1046/j.1540-8167.2003.02500.x. PMID 12741703
- [Background] Link MS, Hill SL, Cliff DL, Swygman CA, Foote CB, Homoud MK, Wang PJ, Estes NA 3rd, Berul CI. Comparison of frequency of complications of implantable cardioverter-defibrillators in children versus adults. Am J Cardiol. 1999 Jan 15;83(2):263-6, A5-6. doi: 10.1016/s0002-9149(98)00834-0. PMID 10073833
- [Derived] Atallah J, Erickson CC, Cecchin F, Dubin AM, Law IH, Cohen MI, Lapage MJ, Cannon BC, Chun TU, Freedenberg V, Gierdalski M, Berul CI; Pediatric and Congenital Electrophysiology Society (PACES). Multi-institutional study of implantable defibrillator lead performance in children and young adults: results of the Pediatric Lead Extractability and Survival Evaluation (PLEASE) study. Circulation. 2013 Jun 18;127(24):2393-402. doi: 10.1161/CIRCULATIONAHA.112.001120. Epub 2013 May 21. PMID 23694966

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thin Leads | Gore PTFE-coated
Started | 525 | 223
Completed | 525 | 223
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thin Leads | Gore PTFE-coated | Total
Number analyzed (Participants) | 525 | 223 | 748
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 384 | 112 | 496
  Between 18 and 65 years | 141 | 111 | 252
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.9 (10.6) | 18.8 (9.6) | 18.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245 | 103 | 348
  Male | 280 | 120 | 400
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 525 | 223 | 748

OUTCOME MEASURES:

1. Primary Outcome: ICD Lead Functionality and Performance by Subtype
Description: Lead survival
Time Frame: 5 years
Population: Intent to compare the survival of thin leads versus PTFE-coated coils.
Measure: Number (95% Confidence Interval); unit: percentage of leads to 5 years
Arm/Group | Thin Leads | Gore PTFE-coated
Number analyzed (Participants) | 525 | 223
percentage of leads to 5 years | 55 [52 to 60] | 92 [88 to 94]

2. Primary Outcome: Compare Ease of Lead Extractability by Subtype
Description: Extraction techniques include simple traction (no locking stylet or sheath) and advanced extraction (locking stylet with a sheath). Compared number of extractions using each technique for single and ePTFE-coated coils.
Time Frame: 5 years
Population: Intent to compare the ease of extraction of isodiametric ICD leads versus ICD leads with PTFE-coated coils.
Measure: Count of Participants; unit: Participants
Arm/Group | Thin Leads | Gore PTFE-coated
Number analyzed (Participants) | 114 | 23
Participants | 53 | 12

3. Secondary Outcome: Number of Patients With Major Complications
Description: Major complications experienced by patients undergoing lead extraction.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Thin Leads | Gore PTFE-coated
Number analyzed (Participants) | 127 | 10
Participants | 3 | 3

4. Secondary Outcome: Comparison of Inappropriate Shocks
Description: Comparison of inappropriate shocks between thin leads and PTFE-coated leads.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Thin Leads | Gore PTFE-coated
Number analyzed (Participants) | 300 | 223
Participants | 33 | 13

ADVERSE EVENTS:
Arm/Group | Thin Leads | Gore PTFE-coated
All-Cause Mortality (participants affected / at risk) | 0/525 | 0/223
Serious Adverse Events (participants affected / at risk) | 5/525 | 1/223
Other Adverse Events (participants affected / at risk) | 39/525 | 14/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thin Leads (N=525) | Gore PTFE-coated (N=223)
Advanced Lead Extraction (Cardiac disorders) | 5 (5) | 1 (1) — Requiring more advanced extraction techniques
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thin Leads (N=525) | Gore PTFE-coated (N=223)
Inappropriate Shocks (Cardiac disorders) | 39 (39) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No